CLINICAL TRIAL: NCT03015103
Title: Safety Dermatological Assessment of Topical Use Product Through Dressings Predictive Studies for Evaluation of Photoirritation and Dermal Photosensitivity
Acronym: SAF DER ASSESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kley Hertz S/A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: Kley Hertz 006
Record Dates: First submitted 2016-12-29; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-12

CONDITIONS: Skin Irritability; Skin Sensitisation

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Experimental group (Experimental): This study is designed as a single group assignment, because the 4 dressings (3 placebos and 1 containing the product) will be applied in all volunteers. This means that the region in which the tested product will be applied will be compared with the other placebo regions in the same volunteer.
  Interventions: Device: Intimate Lubrificant Gel

INTERVENTIONS:
Device: Intimate Lubrificant Gel — All the volunteers will receive the application of four dressings (3 placebos and 1 containing the tested product). After a certain period of time, photoirritation and photosensitization will be measured through the evaluation of tested region.

SUMMARY:
The purpose of this study is to prove the product tested does not cause photoirritation or photosensitization reactions when exposed to sun light.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 70 years old;
* Skin types: I (light caucasian) or III (light brown);
* Intact skin where the product will be applied;
* Agreement to comply with the test procedures and attend the clinic in the days and fixed times for medical assessments and application and reading of dressings
* Signature of informed consent form

Exclusion Criteria:

* Pregnancy and lactation
* Use of anti-inflammatory and immunosuppressive from 30 days up to three months prior to selection;
* Diseases that cause immune suppression;
* Use of photosensitizing drugs;
* History or photodermatoses activities;
* Personal or family history of photoinduced skin cancer;
* Presence of precursor lesions of skin cancer, such as melanocytic nevi and actinic keratoses;
* Intense sun exposure in the experiment area Use of new drugs and/or cosmetics during the experiment;
* Previous participation in a study with the same product under test;
* Relevant medical history or current evidence of alcohol or other drugs abuse;
* Known historical or suspected intolerance to any ingredient of the product under study (product under test or comparator);
* Sponsor's employees involved in the study, or close family member of an employee involved in the study;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Photoirritation as measured through the use of dressings containing tested product and placebo | 5 days
  The photoirritation will be measured with the use of four dressings that will be applied in the volunteer (3 dresssings containing different placebos and 1 containing the product). After some hours, the region is evaluated and radiated with UVA. That procedure occurs during the period of five days.
Photosensitization as measured through the use of dressings containing tested product and placebo | 32 days
  The photosensitization will be measured with the use of four dressings that will be applied in the volunteer (3 dresssings containing different placebos and 1 containing the product). After some hours, the region is evaluated and radiated with UVA. That procedure occurs during the period of 32 days.